CLINICAL TRIAL: NCT06656338
Title: Phase 2 Seattle Dietary Biomarkers Development Center (P2-SDBDC)
Brief Title: Phase 2 Seattle Dietary Biomarkers Development Center
Acronym: P2-SDBDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marian Neuhouser (Other)
Collaborators: United States Department of Agriculture - National Institute of Food and Agriculture (USDA-NIFA) (Unknown); University of Nebraska (Other); University of Washington (Other); Duke University (Other)
Responsible Party: Sponsor-Investigator, Marian Neuhouser, Professor, Cancer Prevention Program Head, Fred Hutchinson Cancer Center
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RG1124404; FHIRB0020415 (Other: Fred Hutchinson Cancer Center Institutional Review Board)
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults
Keywords: Healthy Eating Index-2020; Cross-over trial; Controlled feeding study; Metabolomics

STUDY DESIGN:
Intervention Model Description: Randomized cross-over
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statisticians Laboratory personnel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Higher HEI-2020 diet followed by lower HEI-2020 diet (Experimental)
  Interventions: Other: Higher HEI-2020 diet followed by lower HEI-2020 diet
- Arm 2: Lower HEI-2020 diet followed by higher HEI-2020 diet (Experimental)
  Interventions: Other: Lower HEI-2020 diet followed by higher HEI-2020 diet

INTERVENTIONS:
Other: Higher HEI-2020 diet followed by lower HEI-2020 diet — Controlled feeding study of HEI-2020 diet. Crossover feeding study of two, 7-day feeding periods with higher HEI-2020 and lower HEI-2020 diets completed in random order.
  Arms: Arm 1: Higher HEI-2020 diet followed by lower HEI-2020 diet
Other: Lower HEI-2020 diet followed by higher HEI-2020 diet — Controlled feeding study of HEI-2020 diet. Crossover feeding study of two, 7-day feeding periods with higher HEI-2020 and lower HEI-2020 diets completed in random order.
  Arms: Arm 2: Lower HEI-2020 diet followed by higher HEI-2020 diet

SUMMARY:
The Seattle Dietary Biomarker Development Center (S-DBDC) aims to advance the science of measuring dietary intake by identification and validation of dietary biomarkers that improve upon self-reported diet. To accomplish this mission, the Seattle DBDC will carry out controlled feeding studies in healthy human volunteers. Metabolomics assays will be conducted on blood and urine specimens collected during the feeding studies for biomarker identification. Stool samples will be collected and archived.

DETAILED DESCRIPTION:
The central mission of the Seattle Dietary Biomarker Development Center (DBDC) is to advance the science of measuring complex dietary exposures by rigorous identification and validation of dietary biomarkers that improve upon measurement error-prone self-reported diet. To accomplish this mission, the Seattle DBDC first conducted a Phase 1 study for biomarker discovery; the Phase 1 study is registered and reported in a separate clinicaltrials.gov record (NCT05580653) as the study design differs from Phase 2.

In Phase 2 (registered in this current clinicaltrials.gov record), the Seattle DBDC will conduct a two-period, crossover, controlled feeding trial to evaluate whether the food biomarkers discovered in Phase 1 are detectable within the context of higher and lower Healthy Eating Index (HEI) 2020 diet patterns and to discover metabolomic biomarkers of higher and lower HEI-2020 diet patterns. A total of 30 healthy adults will complete two feeding periods in random order. Each feeding period consists of a 2-day run-in of controlled feeding followed by a 7-day feeding period, with at least a 7-day washout between feeding periods. Metabolomics assays will be conducted on blood and urine specimens collected during the feeding studies for biomarker identification and validation. Stool samples will be collected and archived for future studies.

ELIGIBILITY:
Inclusion criteria:

* Healthy adults;
* Age 18 years or older;
* Willing to come to the Fred Hutch campus 10 times during the study; BMI 18.5-39.9 kg/m2

Exclusion criteria:

* Pregnancy or lactation;
* allergy or aversion to any of the foods that will be studied and/or provided;
* history of gastrointestinal disorders including ulcerative colitis, Crohn's disease, celiac sprue, hereditary non-polyposis colorectal cancer (HNPCC), familial adenomatous polyposis, pancreatic disease, or liver disease;
* previous gastrointestinal resection or bariatric surgery;
* bleeding disorders that precludes blood draws;
* recent hospital admissions (past 6 months) for heart disease (MI/CVA or CHF) or other CVD/CAD conditions under physician guided therapy that is not medically stable;
* cancer under radiation or chemotherapy treatment that is active or within 6 months of treatment;
* weight change (±5% in the last 3 months);
* regular alcohol intake of > 2 drinks/day (equivalent to 720 mL of beer, 240 mL of wine, or 90 mL of spirits), and unwilling to abstain during feeding periods;
* use of tobacco and/or marijuana, hookahs, e-cigarettes (e-cigs, vapes, etc) and not willing to abstain during feeding periods;
* use of illicit drugs and not willing to abstain during feeding periods;
* BMI ≥40 kg/m2; regular (daily to weekly) use of over-the-counter (OTC) weight-loss aids or anti-inflammatories, and unwilling or unable to stop taking these during feeding periods;
* unwilling to stop taking OTC dietary supplements that interfere with the test foods being studied including pills, chewables, liquids or powders for the following: protein supplements, soy, fiber, flaxseed, fish oil (including cod liver oil), probiotics, carotenoids, selenium, other antioxidants, other phytochemicals, glucosamine and chondroitin (if vitamin supplement is MD prescribed - may continue);
* oral or IV antibiotic use in the past 6 months (could defer participation until 6 months post-completion of course of antibiotics);
* seated blood pressure >140/90 mmHg; fasting clinical lab tests outside acceptable values as ascertained at the screening blood draw (see Table 2 in protocol document);
* current use of specific prescription medication(s) (see Table 3 in protocol document); and
* inability to freely give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Plasma metabolite concentration at Day 7 for Higher HEI-2020 Diet | Day 7
Urine metabolite concentration at Day 7 for Higher HEI-2020 Diet | Day 7
Plasma metabolite concentration at Day 7 for Lower HEI-2020 Diet | Day 7
Urine metabolite concentration at Day 7 for Lower HEI-2020 Diet | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Marian L. Neuhouser, PhD, RD, Principal Investigator — Fred Hutchinson Cancer Center; Johanna W. Lampe, PhD, RD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will comply with the NIH Data Sharing Policy. This trial will be registered at ClinicalTrials.gov. We will publish results in peer-reviewed journals. Data generated from this study will be sent to the Data Coordinating Center Center (DCC) at Duke University. The DCC will make study data available to other Consortium members (University of California Davis, Harvard University) in accordance with best practices for data safety and accessibility. Participants' data may be stored and shared for future research without additional informed consent if identifiable private information is removed. Use of participant data may result in commercial profit; however, participants will not be compensated for the use of their data other than what is described in the consent form. The final de-identified study data and results will be made publicly available, in accordance with NIH data sharing policies.
Supporting Information: Study Protocol, SAP, ICF